CLINICAL TRIAL: NCT03360292
Title: Describing the Differences in Oxygen Profiles in Premature Infants of Less Than 29 Weeks Gestational Age When Targeted to an Oxygen Saturation Range 92 to 97%, Compared to 90 to 95%
Brief Title: Measuring Oxygenation of Newborn Infants in Targeted Oxygen Ranges
Acronym: MONITOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AC17098; 194632 (Registry Identifier: IRAS)
Record Dates: First submitted 2017-11-27; First posted 2017-12-04 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2019-09

CONDITIONS: Premature Infant; Hypoxia; Hyperoxia
Keywords: Neonatology
MeSH Terms: conditions — Premature Birth; Hypoxia; Hyperoxia

STUDY DESIGN:
Intervention Model Description: This is a randomised cross-over study of oxygen target ranges in premature infants, with infants acting as their own controls.
Masking Description: Infants will be randomised to either higher (92-97%) or lower (90-95%) oxygen saturation target range, and then cross-over to the alternative range after 6 hours of monitoring (with 12 hours in total study time). The study is randomised but not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Higher target range (Experimental): Infants will be targeted to 92-97% oxygen saturation
  Interventions: Other: Higher target range
- Standard target range (No Intervention): Infants will be targeted to 90-95% oxygen saturation, which is the range used as routine in the Neonatal Unit involved in the study

INTERVENTIONS:
Other: Higher target range — Intervention is using a higher oxygen saturation target range than in routine practice
  Other Names: Using a higher oxygen saturation target range
  Arms: Higher target range

SUMMARY:
The investigators aim to measure the effect of targeting premature babies to a slightly higher oxygen saturation target range (92-97%) than routinely used, for a brief period, to plan a future larger study of the effect of this on clinical outcomes.

It is still unclear exactly what levels of oxygen premature babies need - both too little or too much oxygen in the first weeks after birth may be harmful. Previous studies used saturation monitoring (SpO2), where a small probe shines light through the skin and calculates how much oxygen is carried in the blood. These studies demonstrated using an SpO2 range of 91-95% rather than 85-89% was associated with more babies surviving and fewer babies suffering from a bowel condition called necrotising enterocolitis (NEC). However, targeting oxygen higher increased the number of infants who needed treatment for an eye condition called retinopathy of prematurity (ROP).

It is possible an SpO2 range higher than 91-95% would be associated with even better survival. It is also possible that a higher range might not improve survival but could increase the need for ROP treatment.

Infants born at less than 29 weeks gestation, greater than 48 hours of age and receiving supplementary oxygen would be eligible for inclusion. The study is at the Royal Infirmary of Edinburgh. Total study time is 12 hours for each infant (6 hours at the standard 90-95% range used in our unit, and 6 hours at 92-97%). It is a crossover study with infants acting as their own controls.

Based on previous research the investigators are confident these oxygen levels will not be dangerously high. To provide an additional measure of oxygen the investigators will also use a transcutaneous monitor for the 12 hour study period, which fastens gently to the skin and measures oxygen and carbon dioxide levels on the skin surface.

DETAILED DESCRIPTION:
This study is a single centre randomised crossover study. Infants born at less than 29 weeks gestation, greater than 48 hours of age and receiving supplementary oxygen would be eligible for inclusion. The study is at the Royal Infirmary of Edinburgh. Total study time is 12 hours for each infant (6 hours at the standard 90-95% range used in our unit, and 6 hours at 92-97%). It is a crossover study with infants acting as their own controls.

A complete list of all monitoring that will be carried out is shown below:

1. SpO2 monitoring
2. TcPO2 monitoring
3. Heart rate monitoring (used to validate SpO2 readings as described below)
4. Arterial gas sampling (only if conducted by the direct care team as part of the routine care of the infant will these be recorded. No extra blood samples will be taken as part of the study)

Each infant will be monitored simultaneously with an SpO2 monitor and TcPo2 monitor, with data recording starting from the time the transcutaneous monitor finishes calibrating. SpO2 readings will be downloaded directly from the multiparameter patient monitor. SpO2 will be measured using a Siemens Infinity SC7000 multiparameter monitor. This monitor uses Siemens' Oxisure pulse oximetry technology and Nellcor Oximax saturation probes and incorporates ECG to reduce motion artefact. To reduce the influence of artefact further, data from an infants chest leads (recording heart rate) will also be downloaded. If there is a greater than 10 beats per minute difference between heart rate measured from the pulse oximeter and heart rate measured from the chest leads, SpO2 for that time point will be disregarded.

TcPO2 will be measured using a SenTec Digital Monitoring System with OxiVent sensor. TcPO2 is calculated by dynamic fluorescence quenching which measures oxygen molecules present in the vicinity of a fluorescent dye incorporated within the sensor surface. The sensor is operated at a constant temperature of 43 degrees Celsius. Control of sensor temperature and application duration are designed to meet all applicable standards and this monitoring device is used routinely in many neonatal units, with transcutaneous monitoring part of the monitoring equipment we use in selected infants in our unit and being transported by our local neonatal transport team. Temperature is supervised by two independent circuits, as well as by the monitor firmware.

Transcutaneous data will be transferred contemporaneously to a bedside PC via the proprietary software V-STATS (with V-CareNeT) version 4.01. We will ensure the time on the monitor is synchronised with the time displayed on the electronic patient record system recording SpO2 and heart rate. V-STATS software can identify any spurious spikes in TcPO2 caused by air bubbles and these identified segments of data will be discarded. Artefact has not significantly affected readings during the routine use of this monitor previously on our neonatal unit and with our neonatal transport team. The site of the transcutaneous probe will be rotated on each infant every 2 hours.

SpO2, TcPO2 and heart rate data will be recorded every second. The time of any arterial oxygen samples taken routinely during the study will be recorded from the unit Radiometer ABL800 FLEX blood gas analyser.

ELIGIBILITY:
Inclusion Criteria:

* Infants born at less than 29 weeks gestation
* Infants greater than 48 hours of age
* Infants who are receiving supplementary oxygen

Exclusion Criteria:

* Congenital anomalies that would affect oxygenation (eg. cardiac defects, congenital diaphragmatic hernia)

Ages: 48 Hours to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2020-01-18 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
Incidence of hyperoxia and hypoxia on saturations | 12 hours
  Percentage time spent above an SpO2 of 97% and below an SpO2 of 90% when infants are targeted to an SpO2 range of 92-97% compared to 90-95%

SECONDARY OUTCOMES:
Incidence of hyperoxia and hypoxia on Transcutaneous monitoring | 12 hours
  To discover the percentage time spent above a TcPO2 of 80mmHg and below a TcPO2 of 50mmHg when infants are targeted to an SpO2 range of 92-97% compared to 90-95%
Saturation variability | 12 hours
  To discover the variability in SpO2 (measured by standard deviation) when infants are targeted to an SpO2 range of 92-97% compared to 90-95%
Transcutaneous variability | 12 hours
  To discover the variability in TcPO2 (measured by standard deviation) when infants are targeted to an SpO2 range of 92-97% compared to 90-95%
Characterise PaO2 values within the two oxygen saturation target ranges | 12 hours
  In infants who are undergoing PaO2 measurement as part of their routine care describe the PO2 values observed in the two target ranges
Pooled frequency histogram of SpO2 | 12 hours
  To generate a pooled frequency histogram of percentage time at each SpO2 point between 80 and 100% for infants targeted to an SpO2 range of 92-97% compared to 90-95%
Pooled frequency histogram of TcPO2 | 12 hours
  To generate a pooled frequency histogram of percentage time at a TcPO2 of below 30mmHg, 30-39.9mmHg, 40-49.9mmHg, 50-59.9mmHg, 60-69.9mmHg, 70-79.9mmHg, and 80mmHg and above for infants targeted to an SpO2 range of 92-97% compared to 90-95%

CONTACTS AND LOCATIONS:
Locations (1):
- Neonatal Unit - Royal Infirmary of Edinburgh, Edinburgh, Lothian, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Christie FG, Kelly R, Boardman JP, Stenson BJ. Measuring Oxygenation in Newborn Infants with Targeted Oxygen Ranges (MONITOR): a randomised crossover pilot study. Arch Dis Child Fetal Neonatal Ed. 2023 Nov;108(6):638-642. doi: 10.1136/archdischild-2022-324833. Epub 2023 May 4. PMID 37142388

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/92/NCT03360292/Prot_SAP_000.pdf
  • Informed Consent Form (2017-11-27): https://cdn.clinicaltrials.gov/large-docs/92/NCT03360292/ICF_001.pdf